CLINICAL TRIAL: NCT00083538
Title: UARK 2000-46, A Phase II Study of Tumor Antigen-Pulsed Autologous Dendritic Cell Vaccination Administrated Subcutaneously or Intranodally in Multiple Myeloma Patients
Brief Title: Study of Tumor Antigen-Pulsed Autologous Dendritic Cell Vaccination Administrated Subcutaneously or Intranodally
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Bart Barlogie, MD, PhD, UAMS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2000-46
Record Dates: First submitted 2004-05-25; First posted 2004-05-27 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; DTPACE; Dexamethasone; Thalidomide; Cisplatin; Cytoxan; Doxorubicin; Etoposide; Dendritic Cell Vaccination; Leukapheresis
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Thalidomide; Cisplatin; Doxorubicin; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dexamethasone
Drug: Thalidomide
Drug: Cisplatinum
Drug: Adriamycin
Drug: Cyclophosphamide
Drug: Etoposide

SUMMARY:
The purpose of this study is to determine if vaccination with autologous idiotype- or tumor lysate-pulsed dendritic cells induces the generation of anti-idiotypic and anti-tumor immunologic responses.

DETAILED DESCRIPTION:
This is an experimental treatment that will consist of receiving special white blood cell administrations either underneath the skin or in the lymph nodes. In this protocol, treatment will be given according to the "risk group". If there are certain abnormalities in the chromosomes, the disease is considered to be high risk. High-risk patients will first receive one cycle of chemotherapy with a regimen called DT PACE, after which the white blood cells will be collected. Leukapheresis is a procedure in which blood is removed, white blood cells are saved, and the remaining blood is given back to you. These dendritic cells will then be mixed with your individual myeloma protein and/or cells, and keyhole limpet hemocyanin (KLH) that is necessary for the enhancement of immune response against myeloma antigens. It is hoped that this will cause these cells to interact with and activate T cells, which will then destroy myeloma cells in your body. Half of these white cells will be injected into your lymph nodes (intranodally) and half will be given subcutaneously. High risk patients will receive a chemotherapy regimen called DT PACE.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have confirmed diagnosis of one of the following: Smoldering or indolent multiple myeloma, Multiple myeloma more than 1 year after autologous transplant and with stable disease, or Multiple myeloma with cytogenetic abnormalities
* Patients with secretory IgA or IgG must have purified idiotype protein available and/or tumor cells available, and patients with light chain or non-secretory myeloma must have tumor cells available
* Karnofsky performance score greater than or equal to 60
* ANC greater than or equal to 1,000/microliters, platelet count greater than or equal to 60,000/microliters, and CD4 count greater than or equal to 400/microliters.
* Expected survival of 3 months or more
* 18 years of age and older
* Have given a written consent and been informed about the investigational nature of the study.
* Negative serology for HIV, Hepatitis C, and negative for hepatitis B surface antigen

Exclusion Criteria:

* Patients with CD4 count < 400/microliters, and/or with severely damaged immune functions
* Chemotherapy or other immunosuppressive treatment with steroids, cytoxan, methotrexate within 8 weeks
* Fever or active infection
* Liver function: total bilirubin greater than or equal to 2 x ULN or AST/ALT greater than or equal to 3 x ULN
* Renal function: Patients on dialysis
* Simultaneous treatment with a second investigational drug or biologic agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To determine if vaccination with autologous idiotype- or tumor lysate-pulsed dendritic cells induces the generation of anti-idiotypic and anti-tumor immunologic responses. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Van Rhee Frits, M.D., Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu